CLINICAL TRIAL: NCT05324241
Title: A Proof of Principle Study of the Laxative Properties of Microencapsulated Lipid in Patients Experiencing Constipation Related to Intentional Weight Loss
Brief Title: Laxative Properties of Microencapsulated Lipid (Constipation Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RS21-058
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microencapsulated fat stomach (Experimental): Participants will consume a drink containing 400kcal of microencapsulated fat that will be released in the stomach.
  Interventions: Dietary Supplement: Fat Microcapsules
- Microencapsulated fat intestine (Experimental): Participants will consume a drink containing 400kcal of microencapsulated fat that will be released in the intestine.
  Interventions: Dietary Supplement: Fat Microcapsules

INTERVENTIONS:
Dietary Supplement: Fat Microcapsules — Consumption of a drink that contains microencapsulated fat that will be released either in the stomach or in the distal small intestines.

SUMMARY:
The present study seeks to build on these observations to assess whether in principle, fat containing microcapsules might help patients experiencing constipation in association with weight loss interventions (including GLP-1 analogues or bariatric surgery) to both avoid/treat constipation and simultaneously optimise their ability to feel full during eating. This potential dual action may provide added benefit versus the use of traditional approaches to constipation prophylaxis e.g., lactulose.

DETAILED DESCRIPTION:
Chronic constipation most frequently arises as a functional disorder of at least 3 months duration, the aetiology of which is multifactorial encompassing dietary and lifestyle factors arising in the context of intact colonic motility. Confirmatory clinical diagnosis of chronic constipation under this definition can be made with reference to the Rome IV criteria encompassing assessment of stool frequency, quality, straining etc.

Whilst broadly prevalent across the population, constipation is particularly troublesome in a significant number of patients undergoing interventions for weight loss in obesity, be that dietary, pharmacological or surgical. Calorie restriction per se, which is a common feature of most interventions for obesity necessarily reduces stimulation of colonic motility by impacting the frequency and intensity of colonic mass movements. Moreover, decreases in dietary fibre during food restriction result in debulking of the stool.

Multiple dietary and pharmacological approaches to the management of chronic constipation are available to mitigate the risk of constipation during weight loss and treat it when it becomes manifest. However, these can often be poorly accepted due to gastrointestinal side effects. Interestingly, the potential laxative properties of orlistat, a pancreatic lipase inhibitor-based treatment for morbid obesity have been investigated in off-label studies in the setting of idiopathic chronic constipation and constipation associated with opioid pain medication and anti-psychotic (clozapine) therapy. Mechanism of action in these cases most probably relates to the pro-kinetic and lubricatory effects of the increasing passage of undigested fat to the colon. Based on these case series, the potential for weight loss pharmacotherapy with in-built mitigation of associated constipation becomes an attractive concept.

When digestive and absorptive processes are impeded or moved distally in the small intestine, as can happen with respect to dietary triglycerides during orlistat therapy, satiety gut hormone signal and quantity of food intake are affected. During an ileal infusion of a lipid emulsion, healthy subjects ate a smaller amount compared to control infusions. A study in healthy volunteers in which fat was delivered via a nasal tube to the duodenum, jejunum and ileum found that the ileal treatment had the most pronounced effect on food intake and satiety.

The investigators have used a new food encapsulation technology using natural food grade pea protein, AnaBio©*, to deliver pure oleic acid to the distal small intestine showed significant attenuation of food intake in association with enhancement of enteroendocrine satiety hormone release. The results recorded an increase in the number of bowel motions over the subsequent 24 hours in half of the participants. Subsequently, the investigators showed that ingestion of a smaller 400kcal cargo of microencapsulated oleic acid resulted in decreased hunger and food intake, no increase in the frequency of bowel motion but an increase in stool softness.

Based on the above data the investigators are encouraged to proceed with the present study, the main goal of which is therefore to investigate whether the 400kcal dose of encapsulated fat delivered to the distal small intestine might be a useful supportive therapy in patients engaged in intensive weight loss therapies and experiencing constipation as a consequence.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Engaged in weight loss treatment
* Diagnosis of chronic constipation (Rome IV criteria)1
* Capacity to consent to participate

Exclusion Criteria:

* Substance abuse
* Pregnancy
* Patients who are taking medication for constipation should be on stable doses of medications for constipation for more than 2 weeks. They should neither start nor stop any medication for constipation in the 2 weeks prior to the visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Completed bowel motion | 24 hours
  Proportion of participants reporting a completed bowel motion within 24 hours.

SECONDARY OUTCOMES:
Hunger | 6 hours
  Hunger scores as measured by Visual Analogue Scales, the scale has a score from 0 to 100 with 0 being least hungry and 100 being most hungry.
calories | 6 hours
  Number of calories consumed during an ad libitum meal
Gut hormones | 6 hours
  Gut hormones concentration
Fullness | 6 hours
  Fullness scores as measured by Visual Analogue Scales, the scale has a score from 0 to 100 with 0 being least full and 100 being most full

CONTACTS AND LOCATIONS:
Overall Officials: Carel le Roux, Principal Investigator — University College Dublin
Locations (1):
- Clinical Research Centre, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No